CLINICAL TRIAL: NCT02735811
Title: The Italian Multicentric OBSERVational Registry on Long-term Outcome of ICD Patients (OBSERVO-ICD Registry)
Brief Title: OBSERVational Registry on Long-term Outcome of ICD Patients
Acronym: OBSERVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Pietro Palmisano, MD, Azienda Ospedaliera Cardinale G. Panico
Other Study IDs: OBSERVO
Record Dates: First submitted 2016-04-02; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Cardiomyopathies
Keywords: Implantable defibrillator; Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Assesment of long-term outcome of ICD patients — Evaluation during follow-up of the occurrence of complications related to ICD implantation and of death
  Other Names: Implantable Cardioverter Defibrillator

SUMMARY:
Multicentric, observational, retrospective registry including patients underwent ICD implantation for any indication. The primary aim of the registry is to evaluate the long-term outcome of patients receiving an ICD.

DETAILED DESCRIPTION:
Multicentric, observational, retrospective registry including patients underwent ICD implantation for any indication in the period from 2010 to 2012. The aims of the registry are to evaluate the occurrence of complications related to ICD implantation (including ICD shocks and electrical storm), and the mortality during a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ICD implantation fo any indication;
* age >18 years

Exclusion Criteria:

* life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients underwent ICD implantation from January 2010 to December 2012 for any indication at enrolling hospitals
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Death for any cause | an average of 2 years

SECONDARY OUTCOMES:
Complications related to ICD implantation | an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Palmisano, MD, Principal Investigator — Cardiology Unit - "Card. G. Panico" Hospital - Tricase
Locations (6):
- Italy (6):
  - University Hospital "Umberto I - Lancisi - Salesi", Ancona, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - AO Pugliese-Ciaccio, Catanzaro, Catanzaro
  - "Card. G. Panico" Hospital, Tricase, Lecce
  - Ospedale Maggiore della Carità, Novara, Novara
  - Ospedale San Filippo Neri, Roma, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerra F, Palmisano P, Dell'Era G, Ziacchi M, Ammendola E, Bonelli P, Patani F, Cupido C, Devecchi C, Accogli M, Occhetta E, Santangelo L, Biffi M, Boriani G, Capucci A; Italian Association of Arrhythmology and Cardiac Pacing (AIAC). Implantable cardioverter-defibrillator programming and electrical storm: Results of the OBSERVational registry On long-term outcome of ICD patients (OBSERVO-ICD). Heart Rhythm. 2016 Oct;13(10):1987-92. doi: 10.1016/j.hrthm.2016.06.007. Epub 2016 Jun 9. PMID 27291511